CLINICAL TRIAL: NCT05000749
Title: A Hybrid Effectiveness-Implementation Multisite Trial of a Dialectical Behavior Therapy Skills Group for Veterans at High-Risk for Suicide Attempt
Brief Title: DBT Skills Groups for Veterans at High Risk for Suicide Attempt
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SDR 20-136
Record Dates: First submitted 2021-08-03; First posted 2021-08-11 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Suicide, Attempted
Keywords: suicide, attempted; dialectical behavior therapy; suicide attempt; emotion regulation
MeSH Terms: conditions — Suicide, Attempted; Emotional Regulation

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two study conditions for the duration of the study.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors will be masked to study condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DBT-SG plus VHA treatment as usual (Experimental): Dialectical Behavior Therapy Skills Group (DBT-SG) in addition to VHA treatment as usual. Group is 24 weekly sessions teaching skills in emotion regulation, distress tolerance, interpersonal effectiveness, and mindfulness.
  Interventions: Behavioral: DBT-SG; Behavioral: VHA treatment as usual
- VHA treatment as usual (Active Comparator): VHA treatment as usual for Veterans at risk for suicide attempt
  Interventions: Behavioral: VHA treatment as usual

INTERVENTIONS:
Behavioral: DBT-SG — Dialectical Behavior Therapy Skills Group (DBT-SG) in addition to VHA treatment as usual. Group is 24 weekly sessions teaching skills in emotion regulation, distress tolerance, interpersonal effectiveness, and mindfulness.
  Arms: DBT-SG plus VHA treatment as usual
Behavioral: VHA treatment as usual — VHA treatment as usual for Veterans at risk for suicide attempt

SUMMARY:
Veteran suicide death is a national crisis. Risk factors include emotion dysregulation, which occurs across mental health disorders. Dialectical behavior therapy (DBT) is an evidence-based suicide intervention that targets emotion dysregulation but is resource-intensive and not widely available at VHA. A more efficient evidence-based DBT Skills Group (DBT-SG) is associated with reduced suicidal ideation and emotion dysregulation and likely more feasible to implement at VHA. This is a randomized controlled trial to test whether DBT-SG in addition to VHA treatment-as-usual, compared to only VHA treatment-as-usual, reduces Veteran emotion dysregulation.

DETAILED DESCRIPTION:
This is a randomized controlled trial at four VHA medical centers. Veterans will be randomized to VHA treatment-as-usual or VHA treatment-as-usual plus DBT-SG.

ELIGIBILITY:
Inclusion Criteria:

* Veteran eligible for VHA care at participating site
* two or more suicide attempts in lifetime, with one in past 12 months, on Columbia-Suicide Severity Rating Scale (C-SSRS)
* current suicidal ideation (endorsing a suicidal ideation scale of at least 1 [passive ideation] on C-SSRS
* emotion dysregulation (score 95 or greater on DERS)
* can attend group sessions
* willing to provide contact information for at least one person who can help locate the participant if study staff are unable to contact them (information for three contact persons will be requested; a participant must provide at least one contact person's information to be included in the study)
* access to telephone; if insufficient access to videoteleconference and local facility is using remote procedures for study, willing to request access to VA-provided device

Exclusion Criteria:

* significant cognitive impairment (score < 28 on modified Telephone Interview for Cognitive Status (mTICS)
* inability to read English or communicate in spoken and written English
* plan to move away or be unavailable in the next 18 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2023-04-30 (Actual); Primary Completion 2027-02-26 (Estimated); Study Completion 2027-02-26 (Estimated)

PRIMARY OUTCOMES:
Change in Emotion dysregulation | Up to18 month follow-up
  Emotion dysregulation will be assessed with the Difficulties in Emotion Regulation Scale, a self-report measure. The scale ranges 36-180 with a higher score indicating greater difficulties in emotion regulation.

SECONDARY OUTCOMES:
Coping | Up to 18 month follow-up
  Coping skills will be assessed with the Dialectical Behavior Therapy Ways of Coping Checklist (DBT-WCCL), a self-report measure. The mean score ranges 0-3 with a higher score indicating greater use of coping strategies.
Columbia-Suicide Severity Rating Scale | Up to 18 month follow-up
  The Columbia-Suicide Severity Rating Scale is a widely used interview measure of suicide risk. The number of suicide attempts during 18month follow-up will be reported (range 0 to infinity), with a higher score indicating more suicide attempts.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Decker, PhD, Principal Investigator — VA Connecticut Healthcare System West Haven Campus, West Haven, CT; Steve Martino, PhD, Principal Investigator — VA Connecticut Healthcare System West Haven Campus, West Haven, CT
Locations (5):
- United States (5):
  - VA San Diego Healthcare System, San Diego, CA, San Diego, California
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut
  - James A. Haley Veterans' Hospital, Tampa, FL, Tampa, Florida
  - New Mexico VA Health Care System, Albuquerque, NM, Albuquerque, New Mexico
  - Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No
Study data will include sensitive information about Veteran suicide risk. In consultation with the VACHS Research Office, the investigators elect not to share final data sets for this reason except as required under FOIA. Data will be preserved at VACHS on secure electronic servers behind the VA firewall, and made available for further study or validation by qualified individuals with VA IRB approval. Contact information for the corresponding mPI will be included in publications to facilitate such requests.

REFERENCES:
- [Derived] Decker SE, Kroll-Desrosiers A, Mattocks KM, Aunon FM, Galliford E, DeRycke EC, Doran N, Baird S, Rielage JK, Ridley J, Bannister J, Giovannelli TS, Fuehrlein BS, Shriver C, Spana E, Honsberger M, Demirelli SA, Shest E, Landes SJ, Goodman M, Martino S. Study protocol of a hybrid type 1 effectiveness-implementation multisite trial: Dialectical behavior therapy skills group for Veterans at high-risk for suicide attempt. Contemp Clin Trials. 2025 Apr;151:107828. doi: 10.1016/j.cct.2025.107828. Epub 2025 Feb 7. PMID 39923893
- [Derived] Decker SE, Kroll-Desrosiers A, Mattocks K, Aunon FM, Galliford E, Doran N, Baird S, Rielage JK, Ridley J, Bannister J, Giovannelli TS, Landes SJ, Goodman M, Walker L, DeRycke E, Shriver C, Spana E, Honsberger M, Brown H, Demirelli S, Shest E, Martino S. Mixed-methods formative evaluation of implementing an adapted suicide prevention treatment: Dialectical Behavior Therapy Skills Groups in the Veterans Health Administration. Front Psychiatry. 2024 Nov 25;15:1495102. doi: 10.3389/fpsyt.2024.1495102. eCollection 2024. PMID 39655211